CLINICAL TRIAL: NCT00706303
Title: Glasgow Supported Self-Management Randomised Controlled Trial for Patients With Moderate/ Severe COPD - GSuST
Brief Title: Glasgow Supported Self Management Trial (GSuST)
Acronym: GSuST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: GG&C Primary Care Division, Greater Glasgow & Clyde NHS Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZH/4/246
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; self management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Intervention group (Active Comparator): Supported Self-management. This will consist of fortnightly individual patient sessions at home of approximately 40 minutes for two months, with home visits at a maximum frequency of 6 weeks thereafter for 1 year. Follow up visits will be less structured, and based on the patient's individual agenda as well as reviewing and reinforcing basic self-management messages. Patients will be provided with an individualised self-management plan and symptom diary cards to use as a monitoring aid. Patients will be trained to identify and treat exacerbations associated with purulent sputum with antibiotic and those associated with increased breathlessness, mucoid sputum and/or upper airway symptoms with Prednisolone.
  Interventions: Behavioral: Supported self management training and support
- 2 (No Intervention): Usual care. The control group will receive usual care, as decided by their GP and or hospital consultant, and the patient themselves (e.g., NHS 24 helpline). They will be asked to complete diary cards and receive telephone follow up calls as an attention control, similar to the intervention group.
  Interventions: Behavioral: Supported self management training and support

INTERVENTIONS:
Behavioral: Supported self management training and support — Supported Self-management. This will consist of fortnightly individual patient sessions at home of approximately 40 minutes for two months, with home visits at a maximum frequency of 6 weeks thereafter for 1 year. Further details of the rubric of the initial training sessions are given in Appendix 1 and will use adapted versions of the Bourbeau self-management and education materials. Follow up visits will be less structured, and based on the patient's individual agenda as well as reviewing and reinforcing basic self-management messages. Patients will be provided with an individualised self-management plan and symptom diary cards to use as a monitoring aid. Patients will be trained to identify and treat exacerbations associated with purulent sputum with antibiotic and those associated with increased breathlessness, mucoid sputum and/or upper airway symptoms with Prednisolone.

SUMMARY:
Training patients to alter their own therapy early in the course of a developing exacerbation (self-management) has been shown to improve outcomes in asthma, but there is no good evidence on this for patients with Chronic Obstructive Pulmonary Disease (COPD). Case management, with patients having an identified contact who helps them access care when necessary, has been shown to improve outcomes in recent studies. A combined approach, called supported selfmanagement, may be particularly suitable for this socially and often educationally disadvantaged group of patients.We propose to identify 500 patients at the time of an exacerbation to test this combined strategy in a randomised manner. The primary outcome measure will be readmission to hospital or death due to COPD, important in terms of patient preferences, quality of life and health costs. This will provide important information about intermediate care for COPD patients which should influence service provision within the NHS in Scotland

DETAILED DESCRIPTION:
There have been no randomised controlled trials from UK settings reporting either the effect or the costs of an intensive, individualised case- and self-management intervention for patients with COPD. Given new evidence from other countries (discussed above), we propose that a combined case- and self-management (henceforth referred to as "supported self-management") intervention is most likely to produce measurable benefits from this socially and physically disadvantaged group of patients. Supported self-management involves:

1. Individualised self-management education, delivered in the patient's own home at fortnightly intervals over a two-month period with monthly telephone follow-up. This component of the intervention is based on an intervention shown to be effective in Canada. It is based on the principle of empowering patients to manage their COPD themselves more effectively by improving disease understanding and symptom monitoring, and improving patients' confidence to carry out appropriate action, such as altering therapy early on in the evolution of an exacerbation or initiating contact with a named professional for telephone advice, a home visit or further hospital care (case management) as and when required. We believe home visits are critical to the success of this intervention as this group of breathless and disabled patients often default from clinics and rehabilitation attendance on account of exacerbations or breathlessness.
2. To maintain the impact of self-management training, a named nurse will visit the patient at (a maximum interval of) six-weeks to reinforce self-management messages; this nurse will also be contactable by the patient, as required, prompting an earlier home visit, or GP or hospital attendance as appropriate.

This supported self-management approach (intervention group) will be compared with standard care (control group).

Aim: To address, via a prospective randomised controlled trial in Glasgow, whether supported self-management, in addition to usual care, in patients with moderate to severe COPD has a measurable benefit on patient morbidity and mortality compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* recent hospital admission with exacerbation
* normal cognitive function (MMSE of 9 or 10)

Exclusion Criteria:

* asthma
* LVF
* malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Difference in COPD admission rates and death over one year between patients treated with supported self-management, in addition to usual care, and those treated with usual care alone? | 1 year

SECONDARY OUTCOMES:
Difference in mean St George Respiratory Questionnaire (SGRQ) scores and the proportion of patients achieving a 4-point improvement in SGRQ mean score at 6 months and 1 year between the intervention and control groups? | 1 year
Difference in length of hospital stay (all causes and sub classified by principle diagnosis) | 1 year
Do demographic variables such as age, sex and social class impact on patient ability to self-manage on the basis of recognising and responding appropriately to worsening symptoms? | i year
Can nurse assistants deliver the combined self- and case-management intervention as effectively as staff nurses, measured by analysis of the appropriateness of behavioural changes in response to worsening symptoms? | 1year
Difference in mean NHS costs, anxiety, depression and self-efficacy scores over 1 year between the intervention group and the control group. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Bucknall, MD, Principal Investigator — GG&C NHS Board
Locations (1):
- Greater Glasgow & Clyde NHS Board, Glasgow, United Kingdom

REFERENCES:
- [Derived] Bucknall CE, Miller G, Lloyd SM, Cleland J, McCluskey S, Cotton M, Stevenson RD, Cotton P, McConnachie A. Glasgow supported self-management trial (GSuST) for patients with moderate to severe COPD: randomised controlled trial. BMJ. 2012 Mar 6;344:e1060. doi: 10.1136/bmj.e1060. PMID 22395923